CLINICAL TRIAL: NCT02813460
Title: A Phase 1, Double-blind, Randomized Study to Assess the Taste Profile of Different ALS-008176 Oral Liquid Formulations in Healthy Adult Subjects
Brief Title: Study to Assess the Taste Profile of Different ALS-008176 Oral Liquid Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108168; 64041575RSV1004 (Other: Janssen Research & Development, LLC); 2016-001517-24 (EudraCT Number)
Record Dates: First submitted 2016-06-02; First posted 2016-06-27 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Session 1: Sequence 1 (Experimental): Participants will sequentially receive 5 milliliters (mL) of each 6 ALS-008176 formulations A B F C E D on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 1: Sequence 2 (Experimental): Participants will sequentially receive 5 mL of each 6 ALS-008176 formulations B C A D F E on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 1: Sequence 3 (Experimental): Participants will sequentially receive 5 mL of each 6 ALS-008176 formulations C D B E A F on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 1: Sequence 4 (Experimental): Participants will sequentially receive 5 mL of each 6 ALS-008176 formulations D E C F B A on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 1: Sequence 5 (Experimental): Participants will sequentially receive 5 mL of each 6 ALS-008176 formulations E F D A C B on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 1: Sequence 6 (Experimental): Participants will sequentially receive 5 mL of each 6 ALS-008176 formulations F A E B D C on day 1.
  Interventions: Drug: Formulation A (ALS-008176); Drug: Formulation B (ALS-008176); Drug: Formulation C (ALS-008176); Drug: Formulation D (ALS-008176); Drug: Formulation E (ALS-008176); Drug: Formulation F (ALS-008176)
- Session 2: Sequence 1 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (G1 G2 H3 G3 H2 H1).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)
- Session 2: Sequence 2 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (G2 G3 G1 H1 H3 H2).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)
- Session 2: Sequence 3 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (G3 H1 G2 H2 G1 H3).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)
- Session 2: Sequence 4 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (H1 H2 G3 H3 G2 G1).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)
- Session 2: Sequence 5 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (H2 H3 H1 G1 G3 G2).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)
- Session 2: Sequence 6 (Experimental): Participants will receive 5 mL of two best scoring formulations from Session 1 with 3 varying concentrations of sucralose (H3 G1 H2 G2 H1 G3).
  Interventions: Drug: Formulation G1 (ALS-008176); Drug: Formulation G2 (ALS-008176); Drug: Formulation G3 (ALS-008176); Drug: Formulation H1 (ALS-008176); Drug: Formulation H2 (ALS-008176); Drug: Formulation H3 (ALS-008176)

INTERVENTIONS:
Drug: Formulation A (ALS-008176) — Reference formulation, 60 mg/mL ALS-008176 oral suspension without sweetener/flavor.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation B (ALS-008176) — 60 mg/mL ALS-008176 oral suspension containing 12 mg/mL sucralose.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation C (ALS-008176) — 60 mg/mL ALS-008176 oral suspension containing 4 mg/mL sucralose and strawberry flavor.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation D (ALS-008176) — 60 mg/mL ALS-008176 oral suspension containing 4 mg/mL sucralose and masking flavor and strawberry flavor.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation E (ALS-008176) — 60 mg/mL ALS-008176 oral suspension containing 4 mg/mL sucralose and masking flavor and cream vanille flavor.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation F (ALS-008176) — 60 mg/mL ALS-008176 oral suspension containing 4 mg/mL sucralose and fantasy fruit flavor.
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation G1 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 1 of sucralose (maximum 12 mg/mL) and best flavor 1 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6
Drug: Formulation G2 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 2 of sucralose (maximum 12 mg/mL) and best flavor 1 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6
Drug: Formulation G3 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 3 of sucralose (maximum 12 mg/mL) and best flavor 1 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6
Drug: Formulation H1 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 1 of sucralose (maximum 12 mg/mL) and best flavor 2 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6
Drug: Formulation H2 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 2 of sucralose (maximum 12 mg/mL) and best flavor 2 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6
Drug: Formulation H3 (ALS-008176) — 60 mg/mL ALS-008176 oral suspension with concentration 3 of sucralose (maximum 12 mg/mL) and best flavor 2 from session 1.
  Arms: Session 2: Sequence 1; Session 2: Sequence 2; Session 2: Sequence 3; Session 2: Sequence 4; Session 2: Sequence 5; Session 2: Sequence 6

SUMMARY:
The purpose of this study is to evaluate in a double-blinded fashion the taste and overall acceptability profile of different ALS-008176 oral liquid formulations as compared to the reference formulation (ALS-008176: 60 milligram per milliliters (mg/mL) oral suspension without sweetener/flavor) for pediatric clinical development and commercialization.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a man or woman between 18 and 65 years of age, inclusive, at Screening
* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* A female participant must be of non-childbearing potential, defined as either: 1) Postmenopausal; 2) A postmenopausal state is defined as no menses for at least 12 months without an alternative medical cause and a serum follicle stimulating hormone (FSH) level in the postmenopausal range (more than [>] 40 international units per liter [IU/L] or milli international units per milliliters [mIU/mL]), or 3) Permanently sterile; 4) Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures (without reversal operation), and bilateral oophorectomy
* During the study and for a minimum of one spermatogenesis cycle (defined as approximately 90 days) after receiving the (last dose of) study drug, a male participant 1) who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example, condom with spermicidal foam/gel/film/cream/suppository); 2) who is sexually active with a pregnant woman must use a condom; 3) must agree not to donate sperm
* Female partners of male participants must either be surgically sterilized, postmenopausal or, if of childbearing potential, must agree to use at least one of the following contraceptive methods for 90 days following the final dose of study drug: a nonhormonal intrauterine device with spermicide; contraceptive sponge with spermicide, diaphragm with spermicide, cervical cap with spermicide, or oral, implantable, transdermal, or injectable-hormonal contraceptives
* A female participant must have a negative serum beta human chorionic gonadotropin (beta hCG) pregnancy test at Screening and a negative urine pregnancy test at Day 1 predose
* A female participant must agree not to donate eggs during the study and for at least 90 days after receiving the (last dose of) study drug
* Participant must have a body mass index; weight (kilogram per height square [kg/height^2 [m^2]) between 18.0 and 30.0 kilogram per meter square (kg/m^2)(inclusive) at Screening
* Participant must be non-smokers and/or have not used chewing tobacco for at least 3 months prior to Screening
* Participant must be able to taste and smell normally, to their own opinion, at all times throughout the study duration. Participants who have an impaired sense of taste and/or smell due to any conditions such as allergic rhinitis, common cold or sinusitis are not eligible to take part in or to continue the study
* Participant must be able to read and write

Exclusion Criteria:

* Participant has a mouth pathology including, but not limited to, pain, ulcer, edema, mucosal erosion, gingivitis and/or (dental) abscesses, or receives treatment for oral pathologies or oral treatment for any disease
* Participant has a history of current clinically significant medical illness including Sjogren's syndrome, cardiac arrhythmias or other cardiac disease, pernicious anemia, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant with a history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy diagnosed in previous studies with experimental drugs
* Participant with presence of any febrile illness or symptoms of upper or lower respiratory tract infection in the 14 days before the (first) dose of study drugs
* Participant has a history of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-V) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse (including barbiturates, opiates, cocaine, amphetamines, methadone, benzodiazepines, methamphetamine, tetrahydrocannabinol, phencyclidine, and tricyclic antidepressants) at Screening
* Participant has known allergies, hypersensitivity, or intolerance to ALS-008176 or its excipients
* Participant has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before the planned first dose of study drug
* Participant is a man who plans to father a child while enrolled in this study or within 90 days after the last dose of study drug, or who is unwilling to use acceptable methods of contraception
* Vulnerable participant (example, incarcerated individuals)
* Participant is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator or participant is an employee of Johnson & Johnson
* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Evaluate in a Double-Blinded Fashion the Taste and Overall Acceptability Profile of Different ALS-008176 Oral Liquid Formulations as Compared to the Reference Formulation (ALS-008176: 60 mg/mL Oral Suspension Without Sweetener/Flavor) | Up to 2 hours of study drug administration
  Taste will be assessed using a questionnaire designed for the purpose. The questionnaire will consist of a visual analogue scale to rate 5 items (sweetness, bitterness, aroma type, aroma strength, and smell) as well as overall acceptability.

SECONDARY OUTCOMES:
Number of participants with adverse events and serious adverse events as a measure of safety and tolerability | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Nottingham, United Kingdom